CLINICAL TRIAL: NCT02731482
Title: Short-and Long-term Effects of a Home-based Rehabilitation Program on Functional Capacity, Peripheral Muscle Strength and Quality of Life in Patients With Bronchiectasis: Randomized Controlled Trial
Brief Title: Short-and Long-term Effects of a Home-based Rehabilitation Program in Patients With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Anderson José, PT, PhD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bronchiectasis Rehabilitation
Record Dates: First submitted 2016-03-30; First posted 2016-04-07 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Rehabilitation; Quality of Life; Physiotherapy Specialty
MeSH Terms: conditions — Bronchiectasis | interventions — Sensitivity Training Groups; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training Group (Experimental): Patients with bronchiectasis in home-based pulmonary rehabilitation
  Interventions: Other: Training Group
- Control Group (Active Comparator): Patients with bronchiectasis in usual care and recommendations for performing exercises
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Training Group — Three sessions per week, each lasting 50 minutes, during eight weeks.
  * Aerobic training in stepping training.
  * Resistance training: Three sets of eight repetitions each, in both simultaneous members, using an elastic band. The trained muscles are quadriceps, hamstrings, deltoid and biceps.
  * Once a week, patients will receive a phone call and every two weeks, patients will get a visit of the researcher at his home.
  Other Names: Physical training intervention
  Arms: Training Group
Other: Control Group — * The participants will receive verbal and written information about the importance of physical activity and walk in moderate intensity, at least, three times a week for 30 minutes.
  * Participants will not receive any supervised physical training.
  * Once a week, patients will receive a phone call to provide support and general advice.
  Other Names: Physical activity intervention
  Arms: Control Group

SUMMARY:
This study will investigate the short-and long-term effects of the home-based pulmonary rehabilitation on peripheral muscle strength, functional capacity and quality of life in patients with bronchiectasis. The participants will be randomized into two groups: control group (usual care and recommendations for practice exercise) and training group, that will perform aerobic (stepping training) and resistance training (lower and upper limbs) for eight weeks, three times a week. At baseline, immediately after finishing and after six months the patients will undergo assessments.

DETAILED DESCRIPTION:
Home-based pulmonary rehabilitation (HBPR) has been used in patients with chronic obstructive pulmonary disease, asthma and pulmonary fibrosis. Results from HBPR have been similar to those observe in the outpatient pulmonary rehabilitation such improvement in exercise capacity, symptoms and quality of life. However, HBPR has not yet been investigated in patients with bronchiectasis, a progressive and debilitating disease with a high socioeconomic impact. Objective: To investigate the short-and long-term effects of the home rehabilitation program in peripheral muscle strength, functional capacity and quality of life in patients with bronchiectasis. Methods: Patients diagnosed with bronchiectasis will be recruited from the Obstructive Diseases Outpatient Clinic of the Hospital das Clínicas - Medicine School, University of São Paulo. Participants will be randomized into two groups: control group (usual care and recommendations for performing exercises and respiratory physiotherapy) and training group, that will perform aerobic (stepping training) and resistance training (lower and upper limbs) for eight weeks, three times a week. All patients will receive a phone call once a week and patients allocated to the training group, additionally, will get a home visit every 15 days. At baseline, immediately after finishing and after six months of the HBPR patients will undergo to assessments. Expected results: HBPR will have positive effects on exercise tolerance and quality of life. Also, this study will contribute to future guidelines on the recommendation of HBPR for patients with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis and/or tomographic bronchiectasis Clinically stable (no change in symptoms of dyspnea, in the amount and color of the secretion) Have completed the outpatient pulmonary rehabilitation for more than a year Not engaged in a regular physical activity.

Exclusion Criteria:

Smokers With other lung related diseases (asthma, COPD and cystic fibrosis) Severe cardiovascular diseases Musculoskeletal limitation Unable to perform the tests and the training protocol due desaturation (pulse oxygen saturation ≤ 80%) over the recommended exercise intensity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Distance, in meters, performed in the Incremental Shuttle Walk Test | up to 9 months
  Measurement of functional capacity and exercise tolerance

SECONDARY OUTCOMES:
Time, in seconds, performed in the Endurance Shuttle Walk Test | up to 9 monthsst
  Measurement of functional capacity and exercise tolerance
Number of steps performed in the Incremental Step Test | up to 9 months
  Measurement of functional capacity and exercise tolerance
Physical functioning domain scale in the Quality of Life Questionnaire-Bronchiectasis (QoL-B) | up to 9 months
  Quality of Life Questionnaire
Kilogram-force (kgf) of quadriceps femoris | up to 9 months
  Peripheral Muscle Strength
Number of steps per day, measured by a pedometer | up to 9 months
  Physical activity in daily life

CONTACTS AND LOCATIONS:
Overall Officials: Simone Dal Corso, PT, PhD, Study Director — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jose A, Holland AE, Oliveira CS, Selman JPR, Castro RAS, Athanazio RA, Rached SZ, Cukier A, Stelmach R, Corso SD. Does home-based pulmonary rehabilitation improve functional capacity, peripheral muscle strength and quality of life in patients with bronchiectasis compared to standard care? Braz J Phys Ther. 2017 Nov-Dec;21(6):473-480. doi: 10.1016/j.bjpt.2017.06.021. Epub 2017 Aug 19. PMID 28869119